CLINICAL TRIAL: NCT05986266
Title: Evaluating Efficacy of Intravenous Carbetocin Versus Intramyometrial Injection of Adrenaline in Reducing Blood Loss During Abdominal Myomectomy: A Randomized Controlled Trial
Brief Title: Evaluating Efficacy of Intravenous Carbetocin Versus Intramyometrial Injection of Adrenaline in Reducing Blood Loss
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Egymedicalpedia (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Micheal Hany Monir
Record Dates: First submitted 2023-08-01; First posted 2023-08-14 (Actual); Last update posted 2023-10-17 (Actual); Status verified 2023-10

CONDITIONS: Uterine Fibroid
MeSH Terms: conditions — Leiomyoma | interventions — carbetocin; Epinephrine

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Active Comparator): patients will receive carbetocin, The optimal carbetocin dose(IV or IM) is 100 mcg. The carbetocin group will receive 100 mcg IV carbetocin (Pabal; Ferring Pharmaceuticals) in 10 mL saline solution. The anesthesiologists will administrate carbetocin slowly over 5 minutes (at a rate of 2 mL/min) to maintain hemodynamic stability.
  Interventions: Drug: Carbetocin
- Group B (Experimental): patients will receive adrenalin, infiltration of the serosa and/or myometrium overlying the leiomyoma before uterine incision with a solution composed of 50 ml Bupivacaine HCL 0.25% and 0.5 mg of adrenaline.The anesthesiologist will be informed prior to the injection of the solution to ensure proper monitoring. The solution will be prepared just before the procedure. Before each infiltration, aspiration will be performed to avoid intravascular injection
  Interventions: Drug: Carbetocin

INTERVENTIONS:
Drug: Carbetocin — To compare efficacy of intravenous carbetocin to intramyometrial injection of adrenaline in decreasing intraoperative blood loss and need for blood transfusion during abdominal myomectomy.
  Other Names: Adrenaline

SUMMARY:
Uterine fibroids, affecting 20-50% of all women ,and are benign tumors that arise from myometrial cells of the uterine smooth muscle tissue. Although most are asymptomatic, fibroids can often cause abnormal uterine bleeding, iron deficiency anemia, pelvic pressure symptoms and pain

DETAILED DESCRIPTION:
Women with myomatous uteri have an increased number of blood supply which may cause excessive bleeding during myomectomy. The excessive bleeding may result in blood transfusions and prolonged hospital stays. A variety of methods are used to reduce bleeding during myomectomy including preoperative administration of gonadotropin-releasing hormone (GnRH) agonists, uterine artery tourniquet, vaginal misoprostol, intravenous tranexamic acid, intramyometrial injections of bupivacaine plus adrenaline and vasopressin, chemical dissection with Mesna (sodium-2-mercaptoethanesulfonate), perioperative injection of ascorbic acid, and, recently, carbetocin.

Currently, there are several strategies for the treatment of fibroids. Still, myomectomy, the surgical removal of myomas, is an important treatment option for symptomatic leiomyomas, especially in women who wish to preserve their uteri.This can be accomplished via laparotomy, laparoscopy or hysteroscopy.

Oxytocin is a hormone secreted from the posterior pituitary and exerts its effect on the uterus by producing uterine contractions during labor and delivery. Because of this contractile feature, synthetic oxytocin analogs are used in the treatment of postpartum uterine atony and hemorrhage. Based on its ability to attenuate blood loss, oxytocin has been evaluated in gynecologic procedures, including hysterectomies, myomectomies, and endometrial resections. Although the expression of oxytocin receptors is thought to be strictly related to pregnancy, their presence has been demonstrated in the leiomyomatous uterus.

Carbetocin was first introduced to control postpartum hemorrhage, but its manageability and efficacy soon made it an interesting option for gynecologic surgeons. Given its longer half-life compared with oxytocin and its ample bioavailability, carbetocin could represent a very useful tool during myomectomy, administered either intravenously or intramuscularly Following promising reports on the effectiveness of carbetocin in reducing intraoperative blood loss, hemoglobin drop, and need for postoperative blood transfusions.

Adrenaline is a potent vasoconstrictive agent that has a high risk of cardiovascular effects if an intravascular instillation is performed. The vasoconstrictive effect of adrenaline on tissue lasts longer than that of vasopressin.

Bupivacaine is a local anesthetic that causes vasodilatation at clinical doses, but lower doses appear to cause vasoconstriction. Bupivacaine has shown to have a vasoconstrictive activity in concentrations of ≤ 0.25%, with duration of its action between 4 and 24 h when used for local infiltration. The use of a combination of bupivacaine and low dose of adrenaline in order to minimize the cardiovascular effects of the latest without interfering with the vasoconstrictive effects on haemostasis has been documented.

The myometrial injection of adrenaline plus bupivacaine was one of the evaluated methods showing significantly reduced blood loss and shorter duration of surgery compared to placebo

ELIGIBILITY:
Inclusion Criteria:

* Women aged 25-50 years old.
* Women who will undergo abdominal myomectomy because of symptomatic stage 3-6 fibroids, according to FIGO staging (Laughlin-Tommaso et al., 2017), with the number of myomas not exceeding five based on the preoperative ultrasonography (US).

Exclusion Criteria:

* Women with previous myomectomy.
* Pregnant and postmenopausal women.
* Women with preoperative hemoglobin concentration <10 g/dL,
* women who are candidate for and choosing vaginal or laparoscopic myomectomy.
* History of preoperative embolization or hormone therapy (GnRH analogues), cervical and broad ligament myoma, number of myomas more than five on preoperative US, myoma FIGO stages 1,2,7 and 8 (Munro et al., 2011)
* Patients with allergy or contraindications to carbetocin or epinephrine, such as coronary artery disease, asthma, epilepsy, migraine, kidney, and hepatic disease.

Ages: 25 Months to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 62 (Actual)
Dates: Start 2023-02-01 (Actual); Primary Completion 2023-08-30 (Actual); Study Completion 2023-09-15 (Actual)

PRIMARY OUTCOMES:
Intraoperative and Post operative bleeding(defined as blood loss ≥500 cc) | First 2 hours after abdominal myomectomy
  Compare efficacy of intravenous carbetocin to intramyometrial injection of adrenaline in reducing intraoperative blood loss during abdominal myomectomy Outcome of the study will be measured in terms of assessment of Hemoglobin level and Hematocrit level pre and post operatively.

SECONDARY OUTCOMES:
Side Effects Of the used drugs in the operation | First 24 hours after abdominal myomectomy
  * Need for blood transfusion.
  * Duration of surgery.
  * Operative complications.
  * Post operative adverse effects such as allergy, cardiovascular disorders and pulmonary edema, etc.

CONTACTS AND LOCATIONS:
Overall Officials: Waleed Saber, Professor, Study Chair — Cairo University
Locations (1):
- Faculty of medicine, Cairo University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided